CLINICAL TRIAL: NCT04236219
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled Single Ascending Dose Study of ALLN-346 (Engineered Urate Oxidase)
Brief Title: ALLN-346 Single Ascending Dose (SAD) Study in Healthy Volunteers
Acronym: SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALLN-346-101
Record Dates: First submitted 2020-01-14; First posted 2020-01-22 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2020-06

CONDITIONS: Hyperuricemia
Keywords: hyperuricemia; gout; urate oxidase; uric acid
MeSH Terms: conditions — Hyperuricemia; Gout

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALLN-346 (Experimental): ALLN-346
  Interventions: Drug: ALLN-346
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALLN-346 — ALLN-346 is novel urate oxidase provided as capsules for oral administration. Single ascending doses within 3 sequential cohorts: Cohort A - 3 capsules administered once, Cohort B - 6 capsules administered once and Cohort C - 12 capsules administered as 6 capsules twice on 1 day.
  Other Names: Engineered urate oxidase
  Arms: ALLN-346
Drug: Placebo — Matching placebo capsules for oral administration. Single ascending doses within 3 sequential cohorts: Cohort A - 3 capsules administered once, Cohort B - 6 capsules administered once and Cohort C - 12 capsules administered as 6 capsules twice on 1 day.
  Other Names: Matching placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of ALLN-346 in healthy volunteers, in this first in human, single ascending dose study. ALLN-346 is an enzyme that degrades urate in the gastrointestinal tract.

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind, placebo-controlled single ascending dose study of orally administered ALLN-346. The study will evaluate the safety and tolerability, inflammation and immunogenicity, pharmacokinetics and pharmacodynamics of ALLN-346 in healthy volunteers. The study consists of a Screening Period, a Treatment Period of 3 days, which includes 1 single day of dosing and 3 days of in-house observation, and a safety Follow-up Period through Day 28 following dosing.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Incapable of pregnancy, not nursing, and agrees to use an effective method of contraception; males subjects must agree to abstain from sperm donation
* Good general health as determined by medical history and physical examination
* Normal clinical laboratory test results and ECG

Exclusion Criteria:

* Presence or history of any significant cardiovascular, gastrointestinal, hepatic, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurological, psychiatric disease or history of hyperuricemia
* Any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines
* Positive screen results for drugs of abuse, alcohol, or cotinine or recent history of drug or alcohol abuse
* Clinically significant abnormal findings on physical examination, vital signs or on electrocardiogram (ECG)
* Positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) antibody
* Received treatment with or exposure to an Investigational drug or device within 30 days prior to or during Screening
* Per Investigator judgment, is not an ideal clinical study candidate

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | 28 days
  Number of participants with treatment emergent adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Anti-drug antibody assessment of immune response | 28 days
  Development of anti-drug antibodies (total Immunoglobin levels, mg/dL)
Serum level of ALLN-346 | 48 hours
  Change of serum ALLN-346 level (ng/mL)
Serum ALLN-346 uricase activity level | 48 hours
  Change of serum ALLN-346 activity (ng/mL)
Serum uric acid assessment of pharmacodynamic response | 48 hours
  Change in serum uric acid concentration (mg/dL)
C-reactive protein (CRP) assessment of inflammation response | 48 hours
  Change in CRP blood levels (mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Tosone, MS, Study Director — Allena Pharmaceuticals, Inc
Locations (1):
- Medpace Clinical Pharmacology, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No